CLINICAL TRIAL: NCT06824636
Title: Comparison of Per Kilogram and Nitrogen Balance Calculations for the Prediction of Daily Protein Requirement in Cancer Patients: A Prospective Randomized Controlled Study
Brief Title: Per Kilogram Versus Nitrogen Balance Methods for Daily Protein Requirement in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Altınkaynak, Ass. Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 158299-2019
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Nitrogen Balance; Cancer; Protein Requirement
Keywords: Cancer; Protein; Diet; Physical performance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Per kg (PK) (Active Comparator): Daily protein requirement was determined by PK in the first group and by NBE in the second group. Patients in the PK group received 1.2-1.5 g/kg/day of protein.
  Interventions: Other: a personalized diet plan was prepared according to the calculated requirements of each patient by two expert dietitians
- Nitrogen Balance Equation (NBE) (Active Comparator): Patients in the NBE group were asked to record their food consumption and to collect a 24-hour urine sample on the same day for nitrogen balance calculation. Nitrogen balance was calculated by subtracting the amount of nitrogen excreted daily (urinary urea/2.14 + 3 g excreted in faeces) from the amount of nitrogen intake (24-h protein consumption [g]/6.25). The predicted daily protein requirement in the NBE group was calculated with daily nitrogen loss x 6.25 (g protein).
  Interventions: Other: a personalized diet plan was prepared according to the calculated requirements of each patient by two expert dietitians

INTERVENTIONS:
Other: a personalized diet plan was prepared according to the calculated requirements of each patient by two expert dietitians — Oral enteral nutrition products were added to the diet if the daily calorie and/or protein requirements could not be met by the diet. All of the patients underwent follow-up visits (4th and 8th weeks) after the initial assessment on admission. Each visit (0, 4th and 8th weeks) included screening of the nutritional status and food consumption, and measurements of body mass index (BMI), muscle mass, muscle strength, gait speed, serum albumin and serum C-reactive protein (CRP). Anthropometric measurements, muscle strength, physical performance, and the physical exercise plan were assessed.

SUMMARY:
The goal of this study is to compare the effects of two dietary protein supplementation methods (per kg [PK] vs nitrogen balance equation [NBE]) on nutritional status, muscle strength, lean body mass, physical performance, and dietary compliance in cancer patients.

The main questions it aims to answer are:

Does the PK method improve muscle strength and lean body mass more effectively than the NBE method?

Which method better supports nutritional status and physical performance in cancer patients?

Are there differences in dietary compliance between the two methods?

Researchers will compare the PK method (1.2-1.5 g/kg/day protein) to the NBE method (protein requirements based on nitrogen balance) to evaluate their impact on these outcomes.

Participants will:

Follow a personalized diet plan based on either the PK or NBE method

Attend follow-up visits at weeks 4 and 8 for assessments of BMI, muscle mass, muscle strength, gait speed, serum albumin, and CRP

Engage in moderate aerobic exercise (brisk walking) for at least 30 minutes a day, 5 days a week

DETAILED DESCRIPTION:
Materials and Methods

Study Population: Cancer patients over 18 years of age, who were admitted to the outpatient clinics of Istanbul University, Institute of Oncology, between September 2019 and January 2020, were included. Informed written consent was obtained from all participants prior to the study. Exclusion criteria were: age below 18, inability to feed orally (due to dementia, impaired consciousness, dysphagia, etc.), dialysis dependence, psychiatric and/or eating disorders, and those on home parenteral nutrition.

Malnutrition Risk ScreeningMalnutrition (MN) risk was screened using the Nutritional Risk Screening 2002 (NRS-2002) tool. Patients with an NRS-2002 score ≥3 were considered at risk of malnutrition.

Assessment of Daily Energy and Protein RequirementsDaily energy requirements (DER) were estimated by adding activity and stress factors to the basal energy requirement calculated using the Harris-Benedict equation. The daily protein requirement was determined using the PK method in one group and the NBE method in the other, with a 1:1 allocation ratio. The PK group received 1.2-1.5 g/kg/day of protein. The NBE group recorded their food intake and collected 24-hour urine samples for nitrogen balance calculation. Nitrogen balance was calculated by subtracting daily nitrogen excretion (urinary urea/2.14 + 3 g from feces) from nitrogen intake (24-hour protein consumption [g]/6.25). The predicted daily protein requirement in the NBE group was calculated as daily nitrogen loss x 6.25 (g protein).

Personalized Diet Plan and Follow-UpA personalized diet plan was prepared for all patients according to their calculated requirements by two expert dietitians from Istanbul University, Istanbul Faculty of Medicine, Clinical Nutrition Team. Oral enteral nutrition products were added if dietary intake was insufficient to meet daily calorie and/or protein needs. Follow-up visits were conducted at the 4th and 8th weeks post-admission. Each visit included assessments of nutritional status, food consumption, BMI, muscle mass, muscle strength, gait speed, serum albumin, and C-reactive protein (CRP).

Measurements of Anthropometrics, Muscle Strength, and Physical PerformanceAnthropometric measurements were performed using bioelectrical impedance analysis (BIA) (Tanita MC 780 MA, Japan) to assess body weight, fat-free mass (FFM), fat ratio, total body water (TBW), bone weight, and visceral adiposity index. BMI was calculated as weight in kilograms divided by height in meters squared. Muscle strength (kg) was measured using a handheld dynamometer (Jamar, USA), with three repetitions per hand, and the highest measurement from the dominant hand was used. Gait speed (m/s) was assessed using a 4-meter walk test. All measurements were conducted by two nurses from Istanbul University, Istanbul Faculty of Medicine, Clinical Nutrition Team.

Physical Exercise PlanModerate-intensity aerobic exercise (brisk walking) for at least 30 minutes per day, 5 days a week, was planned for each patient by a physiotherapist from the Physical Therapy and Rehabilitation Department.

ELIGIBILITY:
Inclusion Criteria:

Cancer patients aged over 18 years

Patients admitted to the outpatient clinics of Istanbul University, Institute of Oncology, between September 2019 and January 2020

Exclusion Criteria:

Patients aged below 18 years

Patients unable to feed orally (such as those with dementia, impaired consciousness, dysphagia, etc.)

Dialysis patients

Patients with psychiatric and/or eating disorders

Patients receiving home parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Strength Based on Different Protein Calculation Methods | Baseline and 8 weeks
  Change in muscle strength from baseline to week 8, measured by a handheld dynamometer.
Change in Lean Body Mass Based on Different Protein Calculation Methods | Baseline and 8 weeks
  Change in lean body mass from baseline to week 8, assessed via bioelectrical impedance analysis (BIA).
Change in Nutritional Status Based on Different Protein Calculation Methods | Baseline and 8 weeks
  Improvement in nutritional status, evaluated using NRS-2002 scores from baseline to week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Saka, Professor, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication